CLINICAL TRIAL: NCT06338098
Title: Investigating the Effect of an 8-week Heartfulness Meditation Program on Employee Burnout and Stress at Veterinary Specialty Hospital
Brief Title: Effect of an 8-week Heartfulness Meditation Program on Burnout and Stress at Veterinary Specialty Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heartfulness Institute (Other)
Collaborators: Angell Animal Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HFNVSH.001
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Stress; Burnout, Professional
Keywords: Heartfulness
MeSH Terms: conditions — Burnout, Professional | interventions — Health

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heartfulness Group (Experimental): Participants in the meditation program will be provided with guided meditation and relaxation audio clips to spend approximately 20 minutes per day on the meditation and relaxation activities and participate each week in a 20-30 minutes online meditation webinar with a certified meditation trainer. All meditation and relaxation exercises can be performed in the comfort of your own home or other place of your choosing. The intervention will be entirely online.
  Interventions: Behavioral: 8-week wellness and relaxation meditation program
- Control Group (No Intervention): The control group had no change in their daily routines.

INTERVENTIONS:
Behavioral: 8-week wellness and relaxation meditation program — Heartfulness Meditation program will be provided with guided meditation and relaxation audio clips to spend approximately 20 minutes per day on the meditation and relaxation activities and participate each week in a 20-30 minutes online meditation webinar with a certified meditation trainer. All meditation and relaxation exercises can be performed in the comfort of your own home or other place of your choosing. The intervention will be entirely online.
  Other Names: 8-week Heartfulness Meditation Program
  Arms: Heartfulness Group

SUMMARY:
This quantitative study assesses the effects of meditation and relaxation practices on the reduction of burnout and stress in veterinary care workers. Assessments at baseline will include the Perceived Stress Scale (PSS) and Maslach Burnout Toolkit, and the same questionnaires were collected in Week 8 and Week 16. The Google form questionnaire will ask the participant for their email address. The form will also include a question eliciting interest in participation in the 8-weeks Heartfulness Meditation program. The program will include tools that promote a heart-based nurturing environment focusing on relaxation, and tools to cope with burnout.

DETAILED DESCRIPTION:
The purpose of this research is to investigate the effects of meditation and relaxation practices on the reduction of burnout and stress in veterinary care workers.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18 years
* An employee of MSPCA-Angell Hospital

Exclusion Criteria:

* Experience suicidal ideation
* Diagnosed with manic-depressive disorders
* Diagnosed with post-traumatic stress disorder (PTSD)
* Diagnosed with psychotic disorders, or any other psychiatric conditions requiring treatment

All eligible members are encouraged to check with their healthcare provider before participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Assess the current level of Anxiety | Week 0
  To assess the current level of stress levels through Perceived Stress Scale. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Changes level of Stress | Week 8 and Week 16
  To assess the beneficial impact of Heartfulness program on lowering the Stress. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Assess the current level of Burnout | Week 0
  To assess the current level of burnout levels through Maslach Burnout Toolkit Scale which included Maslach Burnout Inventory for healthcare professionals (MBI-HSS) and Areas of Worklife (AWS). The MBI-HSS comprised 22 questions across 3 subscales; Emotional Exhaustion (EE)-9 questions, Depersonalization (DP)-5 questions, and self-perceived lack of Personal Accomplishment (PA)-8 questions. Responses were scored on a six-point Likert scale (ranging from 0 = never to 6 = everyday) for each subscale, and tabulated into three tiers (low, moderate or high) based on the reference ranges provided with the MBI-HSS. The higher the score the worse the burnout levels. The AWS is a 28 item questionnaire subdivided into six areas with a response scale of 1 (Strongly Disagree) to 5 (Strongly Agree). Higher the score in a sub-area shows a better area in work life.
Changes level of Burnout | Week 8 and Week 16
  To assess the beneficial impact of Heartfulness program on improving burnout levels through Maslach Burnout Toolkit Scale which included Maslach Burnout Inventory for healthcare professionals (MBI-HSS) and Areas of Worklife (AWS). The MBI-HSS comprised 22 questions across 3 subscales; Emotional Exhaustion (EE)-9 questions, Depersonalization (DP)-5 questions, and self-perceived lack of Personal Accomplishment (PA)-8 questions. Responses were scored on a six-point Likert scale (ranging from 0 = never to 6 = everyday) for each subscale, and tabulated into three tiers (low, moderate or high) based on the reference ranges provided with the MBI-HSS. The higher the score the worse the burnout levels. The AWS is a 28 item questionnaire subdivided into six areas with a response scale of 1 (Strongly Disagree) to 5 (Strongly Agree). Higher the score in a sub-area shows a better area in work life.

CONTACTS AND LOCATIONS:
Locations (1):
- Angell Animal Medical Center,, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Publish a research paper with details on the study design, protocol, analysis of data, and report on implications to stress management and wellness tools.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting six months after publication
Access Criteria: Access criteria IPD and any additional supporting information will be shared with the researchers furthering research in stress management and emotional wellness tools.